CLINICAL TRIAL: NCT04900701
Title: The Impact of Energy Intake and Short-term Disuse on Muscle Protein Synthesis Rates and Skeletal Muscle Mass in Middle-aged Adults.
Acronym: PIE
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Exeter (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 201209-B-01
Record Dates: First submitted 2021-05-20; First posted 2021-05-25 (Actual); Last update posted 2025-01-16 (Actual); Status verified 2025-01

CONDITIONS: Muscle Atrophy; Aging; Energy Malnutrition Protein
Keywords: Muscle protein synthesis; Ageing; Dietary protein; Disuse
MeSH Terms: conditions — Muscular Atrophy; Protein-Energy Malnutrition

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Hypocaloric (Experimental): Participants placed in energy restriction.
  Interventions: Other: Energy status
- Energy Balance (Experimental): Participants placed in energy balance.
  Interventions: Other: Energy status
- Hypercaloric (Experimental): Participants placed in energy surplus.
  Interventions: Other: Energy status

INTERVENTIONS:
Other: Energy status — Varying conditions of energy intake, thereby manipulating whether participants are in a state of energy restriction, balance, or surplus.

SUMMARY:
In healthy middle-aged men and women, what is the effect of dietary energy restriction and energy surplus on daily muscle protein synthesis rates and muscle morphology, compared to energy balance, during free-living and immobilisation?

DETAILED DESCRIPTION:
Background Age related muscle tissue loss, which is associated with a number of negative health outcomes is partially caused by blunted muscle protein synthesis rates (MPS) in response to food ingestion, which is exacerbated by muscle disuse. Concomitantly, consuming an energy balanced diet appears to become more challenging with advancing age, due to a reduction in appetite. Of concern is that the impact of energy intake on muscle protein metabolism during ageing is poorly characterised.

Objective To determine daily MPS and muscle morphology in response to differing energy intakes, in free-living conditions and during immobilisation.

Methods Healthy middle-aged volunteers will consume a hypocaloric, energy-balanced, or hypercaloric diet (providing 1.4 g.kg.day protein) over a three-day free-living period, and a three day period of single leg immobilisation. Deuterium oxide and MRI scans will be used to measure daily MPS and muscle size, respectively.

Value The study will determine the effect of energy intake per se on daily muscle protein synthesis rates and muscle size, in free-living and immobilised conditions. This will inform how energy provision modulates tissue loss with ageing, and how this interacts with the catabolic stress of muscle disuse.

ELIGIBILITY:
Inclusion Criteria:

Age 35-65 Healthy Non-smoker Recreationally active

Exclusion Criteria:

Any diagnosed metabolic impairment (e.g. type 1 or 2 Diabetes) Any diagnosed cardiovascular disease or hypertension Elevated blood pressure at the time of screening. (An average systolic blood pressure reading of ≥150mmHg over two or more measurements and an average diastolic blood pressure of ≥90mmHg over two or more measurements.) Chronic use of diabetic medication. A personal or family history of epilepsy, seizures or schizophrenia. Allergic to mycoprotein / Quorn, penicillin, or cow's milk. Any musculoskeletal injury that may impair their use of crutches. Any diagnosed severe digestive illness. Any diagnosed severe autoimmune disease. Any diagnosed cancer. Any metal fragments in the eyes, a pacemaker, or metal implants in the body that preclude MRI scanning.

Ages: 35 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2021-11-01 (Actual); Primary Completion 2024-06-01 (Actual); Study Completion 2025-06 (Estimated)

PRIMARY OUTCOMES:
Muscle protein synthesis (MPS) | 6 days (3 days free-living, 3 days immobilised)
  Daily muscle protein synthesis rates, expressed as fractional synthetic rate (FSR) (%/day)

SECONDARY OUTCOMES:
Muscle morphology. | 3 day immobilisation phase.
  Changes in muscle size, measured via MRI scanning, during immobilisation.

CONTACTS AND LOCATIONS:
Locations (2):
- United Kingdom (2):
  - Sport & Health Sciences University of Exeter, Exeter, Devon
  - University of Exeter, Sports & Health Sciences, College of Life & Environmental Sciences, Exeter, Devon

IPD SHARING:
Plan to Share IPD: No